CLINICAL TRIAL: NCT02346526
Title: A Single-arm Open Label Biomarker Study of Standard-of-care Radium-223 Chloride for Metastatic Castration-resistant Prostate Cancer
Brief Title: A Biomarker Study of Standard-of-care Radium-223 Chloride for Metastatic Castration-resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Philip J. Saylor, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-375; ONC-2013-119 (Other: Bayer)
Record Dates: First submitted 2015-01-13; First posted 2015-01-27 (Estimated); Results first posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Prostate Cancer; Castration-resistant Prostate Cancer; Castration-resistant Prostate Cancer Metastatic to Bone
Keywords: Prostate Cancer; Castration-resistant prostate cancer; Castration-resistant prostate cancer metastatic to bone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Hematologic Tests; radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radium-223 dichloride (Experimental): After the screening procedures confirm that a patient is eligible to participate in the research study.
  Ra-223- Each treatment cycle lasts 4 weeks during which the patient receives Ra-223 by intravenous infusion on day 1 only. Treatments are given every 4 weeks for a total of 6 treatments. These treatments are designed to be entirely standard. Extra testing during and after that six month period will be added to standard testing and monitoring.
  * Blood Tests
  * CT scan
  * Bone scan
  * FACBC PET/MRI in a subset of participants
  Interventions: Procedure: Blood Tests; Procedure: CT scan; Procedure: FACBC PET/MRI in a subset of participants; Drug: Radium-223 dichloride; Procedure: bone scan

INTERVENTIONS:
Procedure: Blood Tests — Blood will be drawn for standard and nonstandard testing on day one, day 4, and weeks 5, 9, 13, 17, 21, 25, 37, and 93.
Procedure: CT scan — Standard CT scans will be carried out prior to treatment, week 9, and week 25.
Procedure: FACBC PET/MRI in a subset of participants — Approximately half of the study patients (n=10) will undergo experimental FACBC PET/MRI testing at 2 time points each: (1) prior to therapy, and (2) week 9.
Drug: Radium-223 dichloride — Ra-223- Each treatment cycle lasts 4 weeks during which the patient receives Ra-223 at a dose of 50 kBq/kg body weight by intravenous infusion on day 1 only. Treatments are given every 4 weeks for a total of 6 treatments.
  Other Names: Xofigo
Procedure: bone scan — Standard bone scans will be carried out prior to treatment, week 9, and week 25.

SUMMARY:
The purpose of this study is to look for markers of how Ra-223 improves the lives of men with prostate cancer. This study makes use of Ra-223 in the standard FDA-approved way, but adds non-standard testing in an attempt to gain insight about how the drug works and how best to track patients who are receiving the drug.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

This research study is designed to examine a treatment strategy that is standard but still relatively new. Ra-223 consists of a series of six infusions given once every 4 weeks. It was FDA approved in 2013 for the treatment of prostate cancer that has spread to bone and has grown despite ADT ("hormonal therapy").

Ra-223 was approved because it was shown to improve the length of the lives of the men with prostate cancer who received it. Despite that important benefit, it is not known to improve other standard markers of prostate cancer such as PSA blood tests (a blood marker that is used to track cancer activity in men who have prostate cancer) and standard imaging scans such as bone scans and computed tomography (CT) scans. If participants and their doctors do not have good markers of whether or not the cancer is responding to therapy, it is harder to make decisions about whether to continue that therapy. This is a current problem.

This study makes use of Ra-223 in the standard FDA-approved way, but adds non-standard testing in an attempt to gain insight about how the drug works and how best to track patients who are receiving the drug.

ELIGIBILITY:
Inclusion Criteria:

* Male age ≥ 18 years.
* Histologically or cytologically confirmed adenocarcinoma of the prostate. Life expectancy of at least 6 months.
* ECOG performance status of zero, one, or two.
* Bone-predominant metastatic CRPC: at least two skeletal metastases on bone scan with no lung, liver, and/or brain metastasis (lymph node metastasis is allowed).
* Symptomatic as defined by either of the following:

  * (a) Regular use of analgesic medication for cancer-related bone pain (≥ level 1; WHO ladder for cancer pain), or
  * (b) Treatment with EBRT for bone pain (though EBRT must be completed ≥12 weeks prior to enrollment in this trial).
* Judged by investigator to have progressive disease sufficient to clinically justify standard-of-care radium-223 treatment.
* Subjects must be able to understand and be willing to sign the written informed consent form.
* All acute toxic effects of any prior treatment have resolved to NCI-CTCAE v4.0 Grade 1 or less at the time of signing the Informed Consent Form (ICF).
* No intention to use cytotoxic chemotherapy within the next 6 months. Subjects must agree to use adequate contraception beginning at the signing of the ICF until at least 6 months after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the principal investigator.
* Acceptable hematology and serum biochemistry screening values:

  * White Blood Cell Count (WBC) ≥ 3,000/mm3
  * Absolute Neutrophil Count (ANC) ≥ 1,500/mm3
  * Platelet (PLT) count ≥ 100,000/mm3
  * Hemoglobin (HGB) ≥10 g/dl (Please note: it is acceptable from the standpoint of study eligibility to undergo transfusion in order to achieve hemoglobin ≥ 10 g/dl)
  * Total bilirubin level ≤ 1.5 x institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
  * Creatinine ≤ 1.5 x ULN
  * Albumin > 25 g/L
* Willing and able to comply with the protocol, including follow-up visits and examinations.

Exclusion Criteria:

* Treatment with cytotoxic chemotherapy within previous 28 days, or failure to recover from AEs due to cytotoxic chemotherapy administered more than 28 days previous (however, ongoing neuropathy is permitted).
* Received any investigational compound within 28 days prior to the first dose of study drug or planned during the treatment period or follow-up.
* Received systemic therapy with radionuclides (e.g., strontium-89, samarium-153, rhenium-186, or rhenium-188, or Radium Ra 223 dichloride) for the treatment of bony metastases.
* Received previous radiotherapy to approximately >25% of bone marrow.
* Other malignancy treated within the last 3 years (except non melanoma skin cancer or low-grade superficial bladder cancer).
* Visceral metastases as assessed by abdominal or pelvic computed tomography (CT) or other imaging modality.
* Presence of brain metastases.
* Lymphadenopathy exceeding 6 cm in short-axis diameter.
* Any size pelvic lymphadenopathy if it is thought to be a contributor to concurrent hydronephrosis.
* Imminent spinal cord compression based on clinical findings and/or magnetic resonance imaging (MRI). Treatment should be completed for spinal cord compression.
* Any other serious illness or medical condition, such as but not limited to:

  * Any infection ≥ National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 Grade 2
  * Cardiac failure New York Heart Association (NYHA) III or IV
  * Crohn's disease or ulcerative colitis
  * Known bone marrow dysplasia
* Fecal incontinence.
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Saylor, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Radium-223 Dichloride: After the screening procedures confirm that a patient is eligible to participate in the research study.
  Ra-223- Each treatment cycle lasts 4 weeks during which the patient receives Ra-223 by intravenous infusion on day 1 only. Treatments are given every 4 weeks for a total of 6 treatments. These treatments are designed to be entirely standard. Extra testing during and after that six month period will be added to standard testing and monitoring.
  * Blood Tests
  * CT scan
  * Bone scan
  * FACBC PET/MRI in a subset of participants
  Blood Tests: Blood will be drawn for standard and nonstandard testing on day one, day 4, and weeks 5, 9, 13, 17, 21, 25, 37, and 93.
  CT scan: Standard CT scans will be carried out prior to treatment, week 9, and week 25.
  FACBC PET/MRI in a subset of participants: Approximately half of the study patients (n=10) will undergo experimental FACBC PET/MRI testing at 2 time points each: (1) prior to therapy, and (2) week 9.
  Radium-223 dichloride: Ra-223- Each treatment cycle lasts 4 weeks during which the patient receives Ra-223 at a dose of 50 kBq/kg body weight by intravenous infusion on day 1 only. Treatments are given every 4 weeks for a total of 6 treatments.
  bone scan: Standard bone scans will be carried out prior to treatment, week 9, and week 25.
Period: Overall Study
Arm/Group | Radium-223 Dichloride
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radium-223 Dichloride
Number analyzed (Participants) | 22
Age, Customized [Median (Full Range); unit: years]
  Age | 71 [49 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 1
  Unknown or Not Reported | 2
Current Use of Bisphosphonates [Count of Participants; unit: Participants] — Bisphosphonates are a group of drugs that work by slowing bone loss.
  Participants
    Yes | 4
    No | 18
Any Prior Use of Docetaxel [Count of Participants; unit: Participants]
  Yes | 5
  No | 17
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status scale describes a participant's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). The ECOG scale ranges from 0 to 5, with lower scores indicating higher levels of functioning.
  Participants
    Score 0 | 10
    Score 1 | 12
    Score greater than or equal to 2 | 0
Extent of disease [Count of Participants; unit: Participants]
  Less than 6 metastases | 8
  6 to 20 metastases | 7
  Greater than 20 metastases | 7

OUTCOME MEASURES:

1. Primary Outcome: Bone Scan Index
Description: Automated bone scan index (aBSI) is an imaging prognostic biomarker used to quantitatively assess effect of therapy. aBSI expresses the tumor burden in bone as a percent of the total skeletal mass. An aBSI value of 1.0 indicates the tumor(s) to be present in 1% of the entire skeleton (arms and legs included).
Time Frame: Baseline to 2 Months
Measure: Mean (Standard Deviation); unit: percentage of skeletal mass
Arm/Group | Radium-223 Dichloride
Number analyzed (Participants) | 22
percentage of skeletal mass
  aBSI at Baseline | 2.90 (3.44)
  aBSI at 2 months | 3.79 (4.28)

2. Secondary Outcome: Percentage of Skeletal Mass Occupied by a Lesion, Stratified by 18 Month Survival Status
Description: Mean change in automated bone scan index (aBSI) at 2 months (i.e. approximately week 9) as assessed by aBSI will be described by 18 month survival status. In other words, decline in aBSI at 2 months on therapy will be evaluated as a predictive biomarker of survival at 18 months.
Time Frame: Baseline and 2 months
Measure: Mean (Standard Deviation); unit: percentage of skeletal mass
Groups:
- Radium-223 Dichloride / Alive at 18 Months; Radium-223 Dichloride / Deceased at 18 Months: After the screening procedures confirm that a patient is eligible to participate in the research study.
  Ra-223- Each treatment cycle lasts 4 weeks during which the patient receives Ra-223 by intravenous infusion on day 1 only. Treatments are given every 4 weeks for a total of 6 treatments. These treatments are designed to be entirely standard. Extra testing during and after that six month period will be added to standard testing and monitoring.
  * Blood Tests
  * CT scan
  * Bone scan
  * FACBC PET/MRI in a subset of participants
  Blood Tests: Blood will be drawn for standard and nonstandard testing on day one, day 4, and weeks 5, 9, 13, 17, 21, 25, 37, and 93.
  CT scan: Standard CT scans will be carried out prior to treatment, week 9, and week 25.
  FACBC PET/MRI in a subset of participants: Approximately half of the study patients (n=10) will undergo experimental FACBC PET/MRI testing at 2 time points each: (1) prior to therapy, and (2) week 9.
  Radium-223 dichloride: Ra-223- Each treatment cycle lasts 4 weeks during which the patient receives Ra-223 at a dose of 50 kBq/kg body weight by intravenous infusion on day 1 only. Treatments are given every 4 weeks for a total of 6 treatments.
  bone scan: Standard bone scans will be carried out prior to treatment, week 9, and week 25.
Arm/Group | Radium-223 Dichloride / Alive at 18 Months | Radium-223 Dichloride / Deceased at 18 Months
Number analyzed (Participants) | 12 | 10
percentage of skeletal mass
  aBSI at Baseline | 1.55 (1.86) | 4.38 (4.25)
  aBSI at 2 months | 2.24 (2.59) | 6.44 (5.60)

3. Secondary Outcome: Circulating Tumor Cell (CTC) Number
Description: The presence of circulating tumor cells (CTCs) in the peripheral blood, will be assessed by by the FDA-approved assay CELLSEARCH® CTC Test, is associated with decreased progression-free survival and decreased overall survival in patients treated for metastatic prostate cancer.
Time Frame: Baseline/Day 1, Day 30, Day 60
Measure: Mean (Standard Deviation); unit: circulating tumor cells
Arm/Group | Radium-223 Dichloride / Alive at 18 Months | Radium-223 Dichloride / Deceased at 18 Months
Number analyzed (Participants) | 12 | 10
circulating tumor cells
  Baseline/Day 1 | 14.70 (29.64) | 18.44 (25.36)
  Day 30 | 24.71 (61.00) | 15.57 (12.37)
  Day 60 | 11.71 (21.51) | 26.86 (28.05)

4. Secondary Outcome: Circulating Biomarkers of the Tumor Microenvironment
Description: Bone turnover markers (i.e., serum bone specific alkaline phosphatase and N-telopeptide) and plasma biomarkers of inflammation and angiogenesis will be assessed serially. Our analyses of circulating biomarkers of the tumor microenvironment were more limited than originally planned due to a freezer malfunction that compromised our frozen samples that had been saved for later batched analyses. The reported values within the table below reflect CTCm score which is a previously described analysis that uses droplet digital PCR to assess gene expression from circulating tumor cells (CTCs) isolated using the microfluidic CTC-iChip. CTCm score, by published convention, does not have units and does not have a normal range.
  In the present study, the normalized CTCm score was calculated as described previously using weighting coefficients. It is considered better to have a lower CTCm score. The table contains [mean (standard deviation)] of CTCm score for each group at the specified timepo
Time Frame: Baseline/Day 1, Day 30, Day 60
Measure: Mean (Standard Deviation); unit: gene expression score per 7.5mL blood
Arm/Group | Radium-223 Dichloride / Alive at 18 Months | Radium-223 Dichloride / Deceased at 18 Months
Number analyzed (Participants) | 12 | 10
gene expression score per 7.5mL blood
  Baseline/Day 1 | 91.11 (201.94) | 302.40 (762.97)
  Day 30 | 102.25 (248.64) | 42.21 (57.95)
  Day 60 | 294.52 (493.61) | 138.29 (138.02)

5. Secondary Outcome: Baseline Pain Score Evaluation as a Predictor of Survival
Description: Pain and narcotic analgesic use was assessed by the 4-item Brief Pain Inventory (BPI). This instrument contains 4 items, with each item reported on a scale of 0-10, meaning that total possible range is 0-40. For each question's 0-10 response scale, 0 meant no pain/interference and 10 meant worst pain imaginable/complete interference.
  Overall survival (OS) was defined as the interval between the start of therapy and the date of death or censor. For the analysis presented in the table, the algorithm of Contal-O'Quigley was applied to the data using leave-one-out jack-knife resampling to determine the optimal division points according to pain score on 4-item BPI at baseline. Each iteration of the algorithm produced an estimate of the "best" division point based on the data. With this method, optimal cut-point for this cohort was baseline total BPI score < 8 vs ≥8. Median survival for each sub-group is reported as months (with range in parentheses).
Time Frame: Baseline through study completion, up to approximately 5 years
Population: Only 20 out of 22 participants were analyzed due to participant non-compliance.
Measure: Median (Full Range); unit: months
Groups:
- Radium-223 Dichloride / Pain Score Greater Than or Equal to 8; Radium-223 Dichloride / Pain Score Less Than 8: After the screening procedures confirm that a patient is eligible to participate in the research study.
  Ra-223- Each treatment cycle lasts 4 weeks during which the patient receives Ra-223 by intravenous infusion on day 1 only. Treatments are given every 4 weeks for a total of 6 treatments. These treatments are designed to be entirely standard. Extra testing during and after that six month period will be added to standard testing and monitoring.
  * Blood Tests
  * CT scan
  * Bone scan
  * FACBC PET/MRI in a subset of participants
  Blood Tests: Blood will be drawn for standard and nonstandard testing on day one, day 4, and weeks 5, 9, 13, 17, 21, 25, 37, and 93.
  CT scan: Standard CT scans will be carried out prior to treatment, week 9, and week 25.
  FACBC PET/MRI in a subset of participants: Approximately half of the study patients (n=10) will undergo experimental FACBC PET/MRI testing at 2 time points each: (1) prior to therapy, and (2) week 9.
  Radium-223 dichloride: Ra-223- Each treatment cycle lasts 4 weeks during which the patient receives Ra-223 at a dose of 50 kBq/kg body weight by intravenous infusion on day 1 only. Treatments are given every 4 weeks for a total of 6 treatments.
  bone scan: Standard bone scans will be carried out prior to treatment, week 9, and week 25.
Arm/Group | Radium-223 Dichloride / Pain Score Greater Than or Equal to 8 | Radium-223 Dichloride / Pain Score Less Than 8
Number analyzed (Participants) | 6 | 14
months | 9.35 [4.10 to 17.50] | 33.85 [2.10 to 49.60]

6. Secondary Outcome: Baseline Global Health Score Evaluation as a Predictor of Survival
Description: Baseline Global Health Score was reported by participants on a scale of 0 ("The worst health you can imagine") to 100 ("The best health you can imagine"). Overall survival (OS) was defined as the interval between the start of therapy and the date of death or censor, expressed here in months.
  For the analysis presented in the table, the algorithm of Contal-O'Quigley was applied to the data using leave-one-out jack- knife resampling to determine the optimal division points according to Global Health Score at baseline. Each iteration of the algorithm produced an estimate of the "best" division point based on the data. With this method, optimal cut-point for this cohort was baseline Global Health Score ≥95 or <95. Median survival for each sub-group is reported as months (with range in parentheses).
Time Frame: Baseline through study completion, up to approximately 5 years.
Population: Only 21 out of 22 participants were analyzed due to participant non-compliance.
Measure: Median (Full Range); unit: months
Groups:
- Radium-223 Dichloride / Global Health Score Greater Than or Equal to 95; Radium-223 Dichloride / Global Health Score Less Than 95: After the screening procedures confirm that a patient is eligible to participate in the research study.
  Ra-223- Each treatment cycle lasts 4 weeks during which the patient receives Ra-223 by intravenous infusion on day 1 only. Treatments are given every 4 weeks for a total of 6 treatments. These treatments are designed to be entirely standard. Extra testing during and after that six month period will be added to standard testing and monitoring.
  * Blood Tests
  * CT scan
  * Bone scan
  * FACBC PET/MRI in a subset of participants
  Blood Tests: Blood will be drawn for standard and nonstandard testing on day one, day 4, and weeks 5, 9, 13, 17, 21, 25, 37, and 93.
  CT scan: Standard CT scans will be carried out prior to treatment, week 9, and week 25.
  FACBC PET/MRI in a subset of participants: Approximately half of the study patients (n=10) will undergo experimental FACBC PET/MRI testing at 2 time points each: (1) prior to therapy, and (2) week 9.
  Radium-223 dichloride: Ra-223- Each treatment cycle lasts 4 weeks during which the patient receives Ra-223 at a dose of 50 kBq/kg body weight by intravenous infusion on day 1 only. Treatments are given every 4 weeks for a total of 6 treatments.
  bone scan: Standard bone scans will be carried out prior to treatment, week 9, and week 25.
Arm/Group | Radium-223 Dichloride / Global Health Score Greater Than or Equal to 95 | Radium-223 Dichloride / Global Health Score Less Than 95
Number analyzed (Participants) | 7 | 14
months | 39.90 [19.30 to 49.60] | 12.85 [2.10 to 33.20]

ADVERSE EVENTS:
Time Frame: through study completion, up to approximately 5 years
Groups:
- Radium-223 Dichloride: Ra-223: Each treatment cycle lasted 4 weeks during which the patient received Ra-223 by intravenous infusion on day 1 only. Treatments were given every 4 weeks for a total of 6 treatments. These treatments were designed to be entirely standard. Extra testing during and after that six month period was added to standard testing and monitoring (blood tests, CT, bone scan, and FACBC (fluciclovine) PET/MRI in a subset of participants).
  Blood Tests: Blood was drawn for standard and nonstandard testing on day 1, day 4, and weeks 5, 9, 13, 17, 21, 25, 37, and 93.
  CT scan: Standard CT scans will be carried out prior to treatment, week 9, and week 25.
  FACBC (fluciclovine) PET/MRI in a subset of participants: Approximately half of the study patients (n=10) underwent experimental FACBC (fluciclovine) PET/MRI testing at 2 time points each: (1) prior to therapy, and (2) week 9. We did not separate the PET/MRI and non-PET/MRI groups within this adverse event reporting because therapy was identical regardless of whether that imaging was done. The PET and MRI used per this protocol were both clinically available tests (i.e., not experimental).
  Radium-223 dichloride: Each treatment cycle lasted 4 weeks during which the patient received Ra-223 at a dose of 50 kBq/kg body weight by intravenous infusion on day 1 only. Treatments were given every 4 weeks for a total of 6 treatments.
  Bone scan: Standard bone scans were carried out prior to treatment, week 9, and week 25.
Arm/Group | Radium-223 Dichloride
All-Cause Mortality (participants affected / at risk) | 18/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 8/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium-223 Dichloride (N=22)
Depression (Psychiatric disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — hand cramp
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — polydipsia
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal and connective tissue disorders - other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — shaking thighs

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT02346526/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT02346526/ICF_001.pdf